CLINICAL TRIAL: NCT06115616
Title: The Impact of Morning Versus Afternoon Aerobic Exercise on Carbohydrate and Lipid Metabolism in Type 1 Diabetes
Brief Title: Morning Versus Afternoon Aerobic Exercise in Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 97516
Record Dates: First submitted 2023-10-23; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Type1diabetes

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exercise
  Interventions: Behavioral: Morning exercise; Behavioral: Afternoon exercise

INTERVENTIONS:
Behavioral: Morning exercise — Exercise before noon in the morning
Behavioral: Afternoon exercise — Exercise in the late after noon

SUMMARY:
Aim. To determine whether the need for exogenous carbohydrate supplementation during exercise in type 1 diabetes is lower during morning exercise compared to afternoon exercise, and whether this is associated with greater lipid oxidation in the morning.

Design and methods Twelve subjects with type 1 diabetes will participate in a randomized crossover study. Subjects will perform moderate intensity at 60% of VO2max for 1 hour during one morning (9 AM) and one afternoon (4 PM). Glucose monitoring will occur every 10 minutes during exercise, and every 5 minutes if blood glucose drops below 3.9 mmol/l. If blood glucose drops below 3.9 mmol/l, glucose infusion will be administered at a rate that keeps blood glucose just above 5 mmol/l. Glucose and palmitate tracers will be infused and indirect calorimetry will be used to assess glucose and lipid metabolism. Blood samples will be gathered to measure tracer levels, growth hormone, cortisol, and free fatty acids (FFA).

Endpoints: Volume of intravenous glucose needed to maintain glucose above 5 mmol/l during the two exercise bouts, lipid- and carbohydrate oxidation rates, time to hypoglycemia, delta blood glucose levels, lipolysis rate, and endogenous glucose production.

DETAILED DESCRIPTION:
Aim. To determine whether the need for exogenous carbohydrate supplementation during exercise in type 1 diabetes is lower during morning exercise compared to afternoon exercise, and whether this is associated with greater lipid oxidation in the morning.

Rationale. Carbohydrate intake requirements to prevent hypoglycemia may vary throughout the day. Determining whether increased carbohydrate requirements are needed in the afternoon will help patients avoid hypoglycemia.

Design and methods Twelve subjects with type 1 diabetes [age 18-65, male/female, >2 years of diabetes duration, multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII))] will participate in a randomized crossover study. Subjects will perform moderate intensity at 60% of VO2max for 1 hour during one morning (9 AM) and one afternoon (4 PM). For both morning and afternoon exercise bouts, subjects will be asked to refrain from exercise for 48hours prior to the test. For the morning exercise bout, the night before subjects will consume a standardized meal at 7 pm, followed by an overnight fast. The afternoon exercise test will be performed 5 hours after an early standardized lunch with full dose of rapid-acting insulin. Basal insulin will be continued in the usual dosage, and starting blood glucose value will be standardized to target 7.0 mmol/l with acceptable range 5.0-9.0 mmol/l prior to initiation of the exercise session. Glucose monitoring will occur every 10 minutes during exercise, and every 5 minutes if blood glucose drops below 3.9 mmol/l. If blood glucose drops below 3.9 mmol/l, an unlabeled glucose infusion will be administered at a rate that keeps blood glucose just above 5 mmol/l.

Glucose and palmitate tracers will be infused to determine differences in diurnal glucose and lipid metabolism during exercise. Indirect calorimetry will be used to measure glucose and lipid oxidation rates. Blood samples will be gathered to measure tracer levels, growth hormone, cortisol, and free fatty acids (FFA) pre-exercise, during exercise, and post-exercise. Continuous glucose monitoring (CGM) and accelerometer activity and sleep data will be collected 24 hours before exercise and for 24 hours after the exercise bout.

Endpoints. The primary endpoint will be the volume of intravenous glucose (g of glucose) needed to maintain glucose above 5 mmol/l during the two exercise bouts. The secondary endpoints will be Lipid- and carbohydrate oxidation rates, time to hypoglycemia, delta blood glucose levels, lipolysis rate, and endogenous glucose production.

Sample size. A sample size of 12 subjects was chosen by use of power calculations based on alike previous studies, and based on clinical observations of carbohydrate requirements during morning and afternoon exercise (expected difference in carbohydrate supplementation of 20 g with a standard deviation of 15 g).

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* male/female
* >2 years of type 1diabetes duration
* multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII)
* physically active

Exclusion Criteria:

* heart conditions
* unawareness
* severe complications to diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * age 18-65
  * male/female
  * >2 years of type 1 diabetes duration
  * multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII)
  * physically active
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
g of glucose | 4 hours
  The primary endpoint will be the volume of intravenous glucose (g of glucose) needed to maintain glucose above 5 mmol/l during the two exercise bouts. During the study day, blood glucose is monitored 2 hours prior to the exercise bout, during the 1 hour exercise bout and 1 hour after the exercise bout. If blood glucose drops below 3.9 mmol/l, glucose infusion is initiated to keep blood glucose just above 5 mmol/l and volume of iv glucose (translated to g of glucose) is recorded. This is done during the 2 study days, and these study days are held 1-3 weeks apart.